CLINICAL TRIAL: NCT06426459
Title: Positive and Negative Effects of Social Media Usage in Adolescent Girls
Brief Title: Social Media Usage in Adolescent Girls
Status: Not yet recruiting | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: German Research Foundation (Other); University Hospital Tuebingen (Other); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: IRTG_P09
Record Dates: First submitted 2024-04-14; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Menstrual Cycle; Oral Contraceptive
Keywords: Social media use; Adolescent girls; Menstrual cycle; Oral contraceptive; Neuroimaging; Women's mental health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood collection for hormonal assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural menstrual cycle: Adolescent girls who have a natural menstrual cycle and have not used any kind of hormonal contraception for at least 6 months.
- Oral contraceptive: Adolescent girls who use combined oral contraceptives for at least 4 months.

SUMMARY:
The study aims to explore the effects of hormonal fluctuations throughout the menstrual cycle on social media use, brain architecture, neural reward processing and reward behavior, and affective status in adolescent girls. Additionally, it strives to compare the effects of exogenous and endogenous hormones on the above-mentioned aspects. For this purpose, the investigators will compare two main groups in the study: 1. Naturally cycling adolescent girls, 2. Adolescent girls using combined oral contraceptives. This study will combine self-report data via questionnaires, ecological data via Ecological Momentary Assessment (EMA), endocrine data via blood collection, and neural data via fMRI assessment to enhance the understanding of the neurobiological mechanisms underlying social media use in adolescent girls. Furthermore, it seeks to elucidate whether there are vulnerable periods throughout the menstrual cycle when adolescent girls are especially prone to dysfunctional social media use and help to design more specific interventions as well as therapy.

DETAILED DESCRIPTION:
For each participant, there is a screening session, a month-long EMA assessment and two experimental fMRI sessions are planned.

After making sure the participants fill the inclusion and exclusion criteria, the investigators will invite them to the laboratory for a screening session (T0). In this session, the participants will provide written informed consent and assent in case of those under 18 years old and written, informed consent for those who are 18 year old. Furthermore, the participants will participate in a standardized clinical interview to screen for mental disorders (Kinder-DIPS). Subsequently, they will be informed about the study details. Finally, they will fill out questionnaires about personality, depressive symptoms, anxiety symptoms, gender identity and norms, mood, loneliness, social media disorder, internet use, social support, and fear of missing out.

Naturally cycling adolescent girls will join the two fMRI measurements (T1 & T2) during the follicular and luteal phase of the menstrual cycle. Adolescent girls using combined oral contraceptives will join the first fMRI measurement during the pill intake period, and the second measurement during the break period. The fMRI sessions will comprise of filling out questionnaires, fMRI measurements, and blood collection for hormonal assessment.

Questionnaires on depressive symptoms, state anxiety, mood, gender identity, self-esteem, loneliness, fear of missing out (FOMO), social media disorder, internet use, social support and social media use will be administered through RedCap platform. This will ensure the assessment of subjective, self-report data and its changes throughout the measurement time of one month.

The sequence of fMRI measurements incudes four main parts, namely anatomical scan, resting-state scan, Effort Allocation Task (EAT), and diffusion tensor imaging (DTI). This protocol ensures the acquisition of the structural and functional data of the brain in the participants. The detailed protocol components are as follows:

1. Anatomical scan: This first sequence of the protocol ensures assessment and insight into the anatomy of the brain, thus providing structural data of the participants' brain. This will last approximately 8 minutes.
2. Resting-state scan: The next sequence involves participants watching a movie that was designed to improve imaging at rest for approximately 10 minutes. This sequence ensures insight into brain activity when no task is being performed and when the participant is at rest.
3. Effort Allocation Task (EAT): This next sequence aims to assess reward processing and reward behavior in the participants. During this task, participants have to exert physical effort on a grip force device when faced with monetary points at stake. There are two types of reward a participant can face; low and high reward. Additionally, there are two difficulty levels during the task, one being easier and the other more difficult. The payoff for the invested effort will be proportional to its duration. The task will last approximately 17 minutes.
4. Diffusion Tensor Imaging (DTI): During the final sequence, participants will undergo DTI assessment to ensure insight into white matter microstructure and connectivity. This will last approximately 7-8 minutes.

To thoroughly investigate the participants' experiences in their natural environments, Ecological Momentary Assessment (EMA) will be conducted. This will be done through an app called m-Path where participants will fill out daily questionnaires about social media use, self-esteem, premenstrual symptoms, and mood throughout one month. A daily questionnaire lasts approximately 10 minutes. This assessment will ensure data about subjective experiences with high ecological validity.

ELIGIBILITY:
Inclusion Criteria:

* Between 15 and 18 years old adolescent girls
* Body mass index(18-25kg/m2)
* Natural menstrual cycle (between 25 to 31 days) OR use of combined oral contraceptives for at least 4 months
* Social media use (e.g., Instagram, TikTok, Snapchat, Facebook, X, BeReal)
* Non-smoking
* German language fluency
* Attending age-appropriate school

Exclusion Criteria:

* Any neurological or psychiatric disease based on the standardized diagnostic interview (Kinder-DIPS)
* Medical problems such as hormonal, metabolic, developmental or chronic diseases (e.g., congenital disorders, diabetes, dysfunctions of the thyroid, or congestive heart failure)
* Pregnancy
* Females who gave birth or were breastfeeding within the last year
* Use of any other kind of steroid hormonal treatment (except combined oral contraceptives) or psychotropic treatment in the last three months
* Females with premenstrual dysphoric disorder(PMDD)
* Not willing to be informed about incidental fMRI findings

Additional exclusion criteria for fMRI:

* Individuals with non-removable metal objects on or in the body such as cardiac pacemaker, artificial heart valve, metal prostheses, metal implants, metal splinters, etc.
* Tattoos (if fMRI-incompatible according to expert guidelines)
* Claustrophobia
* Surgery less than three months ago
* Pathological hearing or increased sensitivity to loud noises
* Neurological disease or injury
* Moderate or severe head injury
* Restricted (corrected) vision

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study participants will be primarily recruited from residents of Tübingen and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-29 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Brain disparities: Contrasting naturally cycling adolescent girls with those using combined oral contraceptives | Measured twice appr. 2-3 weeks apart; approximately 45 minutes each time
  Possible differences between naturally cycling adolescent girls and those taking combined oral contraceptives in brain structure
Brain disparities: Contrasting naturally cycling adolescent girls with those using combined oral contraceptives | Measured twice appr. 2-3 weeks apart; approximately 45 minutes each time]
  Possible differences between naturally cycling adolescent girls and those taking combined oral contraceptives in brain function (functional activation based on BOLD effect)
Reward-processing disparities: Contrasting naturally cycling adolescent girls with those using combined oral contraceptives | Measured twice appr. 2-3 weeks apart; approx. 17 minutes each time
  Possible differences between naturally cycling adolescent girls and those taking combined oral contraceptives on reward processing
Social media use disparities: Contrasting naturally cycling adolescent girls and those using combined oral contraceptives | Measured through ecological momentary assessment every day throughout one month
  Possible differences in social media use between the two groups

SECONDARY OUTCOMES:
Social media use disparities: Contrasting follicular and luteal phase in naturally cycling adolescent girls | Measured through ecological momentary assessment every day throughout one month
  Possible differences between the two phases of the menstrual cycle in social media use
Brain Disparities: Contrasting follicular and luteal phase in naturally cycling adolescent girls | Measured twice appr. 2-3 weeks apart; circa 45 minutes each time
  Possible differences in brain function and structure in naturally cycling girls in follicular vs. luteal phase
Reward-processing disparities: Contrasting follicular and luteal phase in naturally cycling adolescent girls | Measured twice appr. 2-3 weeks apart; circa 45 minutes each time
  Possible differences in reward processing and reward behavior between the two menstrual cycle phases
Associations between personality and brain function & structure | Measured twice appr. 2-3 weeks apart; circa 45 minutes each time
  Possible effects of personality type on brain structure and brain function for both groups. Personality measured by the NEO-Five-Factor-Inventory.
Associations between personality and reward processing & behavior | Measured twice appr. 2-3 weeks apart; circa 17 minutes each time
  Possible effects of personality type on reward processing for both groups. Personality measured by the NEO-Five-Factor-Inventory.
Self-esteem differences: Contrasting follicular and luteal phase in naturally cycling adolescent girls | Measured through ecological momentary assessment every day throughout one month
  Possible differences in self-esteem between the two phases of the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Renner, Prof. Dr. med., Principal Investigator — Child Psychiatry, University Clinic Tübingen; Tomas Furmark, Dr., Principal Investigator — Department of Psychology, Uppsala University, Sweden
Locations (1):
- University Clinic Tuebingen, Department of Psychiatry & Psychotherapy, Tübingen, Baden-Wurttemberg, Germany